CLINICAL TRIAL: NCT00903006
Title: A Phase I-II, Randomization, Open-Label Clinical Trial of Fulvestrant Versus the Combination of Fulvestrant, MK-0646, and Dasatinib as First-Line Therapy for Metastatic Hormone Receptor-Positive HER2-Negative Breast Cancer
Brief Title: Trial of Fulvestrant, MK-0646, and Dasatinib for Metastatic Hormone Receptor-Positive HER2-Negative Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Merck Sharp & Dohme LLC (Industry); Commonwealth Foundation for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0336
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Breast; Hormone receptor-positive metastatic breast cancer; Fulvestrant; Faslodex; MK-0646; Dasatinib; BMS-354825; Sprycel; Adjuvant hormonal therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; dalotuzumab; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Fulvestrant (Active Comparator): Group 1 will receive Fulvestrant only.
  Interventions: Drug: Fulvestrant
- Group 2: Fulvestrant + Dasatinib (Active Comparator): Group 2 will receive Fulvestrant and Dasatinib.
  Interventions: Drug: Fulvestrant; Drug: Dasatinib
- Group 3: Fulvestrant + MK-0646 (Active Comparator): Group 3 will receive Fulvestrant and MK-0646.
  Interventions: Drug: Fulvestrant; Drug: MK-0646
- Group 4: Fulvestrant, MK-0646 + Dasatinib (Active Comparator): Group 4 will receive Fulvestrant, MK-0646, and Dasatinib.
  Interventions: Drug: Fulvestrant; Drug: MK-0646; Drug: Dasatinib

INTERVENTIONS:
Drug: Fulvestrant — Starting dose of 500 mg through a needle into muscle on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 and beyond. On Day 1 of Cycle 1, injections into 2 different muscles, all other times one injection.
  Other Names: Faslodex
Drug: MK-0646 — Group 3 or Group 4, receive starting dose of 5 mg/kg by vein on Days 1, 18, 15, and 22 of every cycle.
  Arms: Group 3: Fulvestrant + MK-0646; Group 4: Fulvestrant, MK-0646 + Dasatinib
Drug: Dasatinib — Group 2 or Group 4, starting dose of 70 mg (capsules) by mouth daily.
  Other Names: BMS-354825; Sprycel
  Arms: Group 2: Fulvestrant + Dasatinib; Group 4: Fulvestrant, MK-0646 + Dasatinib

SUMMARY:
The goals of this clinical research study are to learn the tolerable and effective doses of the drug MK-0646 that can be given in combination with Sprycel (dasatinib) and Faslodex (fulvestrant) to patients with hormone receptor-positive metastatic breast cancer. The safety of these drugs will be studied as well as markers in the tumors that may help researchers predict the tumors' reaction to the treatment.

DETAILED DESCRIPTION:
The Study Drugs:

Fulvestrant is designed to block estrogen from helping breast cancer tumor cells grow. By blocking estrogen, it may stop tumor growth.

Dasatinib is designed to change the function of genes. By changing the function of these genes, it may prevent cancer from growing and spreading.

MK-0646 is designed to block proteins that help breast cancer cells grow. By blocking these proteins, it may cause the cancer cells to die.

Study Procedures:

You will have a fine needle aspiration or core needle biopsy before you start the study treatment and after 2 weeks. These biopsies are to study genes and proteins, and to see how they change with treatment.

Study Groups:

If you are found to be eligible to take part in this study: you will be enrolled in Phase I or Phase II of the study, depending on when you join the study.

If you are in Phase I, you will be assigned to either Group 1, 2, 3, or 4. If you are in Phase II, (based on the result of the screening biopsy) you will be randomly assigned (as in a roll of dice) to either Group 1, 2, 3, or 4:

* Group 1 will receive fulvestrant only.
* Group 2 will receive fulvestrant and dasatinib.
* Group 3 will receive fulvestrant and MK-0646.
* Group 4 will receive fulvestrant, MK-0646, and dasatinib.

All participants will receive the same dose level of fulvestrant.

If you are in Groups 2, 3, or 4, the dose of MK-0646 and/or dasatinib you receive will depend on when you joined this study. The first set of participants in each group will receive the lowest dose level of MK-0646 and/or dasatinib. Each new set will receive a higher dose of MK-0646 and/or dasatinib than the set before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of MK-0646 and/or dasatinib is found. This is called the Phase I portion of the study.

If you are enrolled in the Phase II portion of the study, you will receive dasatinib at the dose that was tolerated in the Phase I portion.

Study Drug Administration:

Every 28 days makes up 1 study cycle.

You will receive fulvestrant through a needle into your muscle on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2 and beyond. You will have 2 injections each time into 2 different muscles.

If you are in Group 3 or Group 4, you will receive MK-0646 through a needle in your vein weekly.

If you are in Group 2 or Group 4, you will take capsules of dasatinib by mouth every day while you are on study. You should take the drug at about the same time each day with a cup (8 ounces) of water. The study staff will give you a card on which you must record every time that you take dasatinib.

Study Visits:

On Day 1 of every cycle for the first 4 cycles, and then every 3 cycles, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking.
* Blood (about 1 tablespoon) will be drawn for routine tests and to see how your immune system may be responding to the study drug.

On Day 1 of each cycle, the following procedure will be performed:

-You will be asked about any side effects you may be having.

On Day 1 of Cycle 1, your vital signs will be measured.

On Days 8 and 22 of Cycle 1, your vital signs and weight will be measured. You will have an ECG.

On Day 15 of Cycle 1, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* You will have an ECG.
* You will have a PET scan
* You will have a core needle biopsy (which removes more tissue) and/or a fine needle aspiration (which has a smaller needle).

On Days 1, 8, 15, and 22 of Cycles 2 and beyond, your weight will be measured.

On Day 1 of Cycle 4 and every 3 cycles after that, you will have CT scans of the chest, abdomen and/or pelvis, to check the status of the disease. If the disease has spread, you may also have a bone scan and/or x-rays of the bones.

If you are taking warfarin to prevent abnormal blood clotting, blood (about 1-2 teaspoons) will be drawn to check your blood clotting function at least 1 time a week until your blood clotting function becomes stable. After that, blood (about 1-2 teaspoons) will continue being drawn to check your blood clotting function as often as the doctor decides is needed.

Length of Study:

You may receive the study therapy until either you experience intolerable side effects or if the disease gets worse; then you will be taken off study.

End-of-Study Visit:

After you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any other drugs you may be taking and about any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be collected for routine tests.
* You will have a hearing test if you received MK-0646.

Four (4), 8, and 12 weeks after the last dose of study drug, blood (about 1 tablespoon) will be drawn to see how your immune system may have responded to the study drug.

This is an investigational study. MK-0646 is not FDA-approved or commercially available. At this time, MK-0646 is only being used in research. Fulvestrant is currently FDA -approved and commercially available for the treatment of metastatic breast cancer in post-menopausal women. Dasatinib is FDA-approved and commercially available to treat chronic myeloid leukemia. At this time, the use of dasatinib in breast cancer patients is investigational.

Up to 40 patients will take part in this study at University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. For the Phase I: Patients with histologically or cytologically confirmed diagnosis of metastatic hormone receptor-positive HER2-negative breast cancer who have received up to one line of endocrine therapy for metastatic disease.
2. Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) or evaluable disease (e.g., bone metastasis, or lesions which do not fulfill RECIST criteria for metastatic disease)
3. Age >/= 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 2
5. Required laboratory values: Absolute neutrophil count (ANC)>/= 1500 cells/mm^3, platelet count >/= 100,000 cells/mm^3, hemoglobin >/= 9 gm/L; bilirubin </= 1.5 * upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 2.5 * ULN; serum creatinine </= 2.0 * ULN
6. Ability to understand the requirements of the study, provided written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments.
7. Patients must be postmenopausal (> 12 months of amenorrhea, bilateral oophorectomy).
8. Patients must have received prior anti-estrogen therapy in the adjuvant setting.
9. Patients may have easily accessible tumors for biopsy (confirmed by interventional radiology).
10. Patients must consent to biopsies.
11. For the Phase II: Patients with histologically or cytologically confirmed diagnosis of metastatic hormone receptor-positive, HER2-negative, breast cancer who have received up to one line of endocrine therapy for metastatic disease.
12. Measurable disease by RECIST or evaluable disease (e.g., bone metastasis, or lesions which do not fulfill RECIST criteria for metastatic disease)
13. Age >/= 18 years
14. ECOG performance status of </= 2
15. Required Laboratory Values: ANC >/= 1500 cells/mm^3, platelet count >/= 100,000 cells/mm^3, hemoglobin >/= 9 gm/L, Bilirubin </= 1.5 * ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 2.5 * ULN
16. Serum creatinine </= 2.0 * ULN
17. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments.
18. Patients must be postmenopausal (> 12 months of amenorrhea, bilateral oophorectomy).
19. Patients must have received prior anti-estrogen therapy in the adjuvant setting.
20. Patients may have easily accessible tumors for biopsy (confirmed by interventional radiology).
21. Patients must consent to biopsies.

Exclusion Criteria:

1. For the Phase I: History of prior malignancies within the past 5 years with the exception of curatively treated basal or squamous cell carcinomas of the skin or carcinoma in situ of the cervix
2. Concurrent severe or uncontrolled medical disease (i.e., systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure, ongoing or recent gastrointestinal bleed, hepatic or cardiac compromise, hypocalcemia, or known platelet function abnormality).
3. Concomitant medication known to prolong QT interval, unless discontinued >/= 7 days of starting dasatinib therapy.
4. Newly diagnosed (within 3 months before enrollment) or poorly controlled (defined as a fasting serum glucose > 160 mg/dl or hemoglobin A1c > 8% at screening), type 1 or 2 diabetes mellitus.
5. Active or untreated brain metastasis
6. Pleural or pericardial effusion of any grade
7. Bone only metastases
8. Patients for whom endocrine therapy is not appropriate (i.e. life threatening metastatic disease).
9. Patients requiring therapeutic anticoagulation (Warfarin 1 mg for port maintenance is allowed).
10. For the Phase II: History of prior malignancies within the past 5 years with the exception of curatively treated basal or squamous cell carcinomas of the skin or carcinoma in situ of the cervix
11. Concurrent severe or uncontrolled medical disease (i.e., systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure, ongoing or recent gastrointestinal bleed, hepatic or cardiac compromise, hypocalcemia, or known platelet function abnormality).
12. Concomitant medication known to prolong QT interval, unless discontinued >/= 7 days of starting dasatinib therapy.
13. Newly diagnosed (within 3 months before enrollment) or poorly controlled (defined as a fasting serum glucose > 160 mg/dl or hemoglobin A1c > 8% at screening), type 1 or 2 diabetes mellitus.
14. Active or untreated brain metastasis
15. Pleural or pericardial effusion of any grade
16. Bone only metastases
17. Patients for whom endocrine therapy is not appropriate (i.e. life threatening metastatic disease).
18. Patients requiring therapeutic anticoagulation (Warfarin 1 mg for port maintenance is allowed).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gonzalez-Angulo, MD, MS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 19, 2009 to February 13, 2012. All recruitment done in medical clinical at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Out of 11 participants registered to the trial, five (5) were screen failures and thus excluded from the trial. The Phase I portion of study began with the first three arms: 1) Fulvestrant, 2) Fulvestrant + Low Dose Dasatinib and 3) Fulvestrant + Low Dose of MK-0646.
Period: Overall Study
Arm/Group | Group 1: Fulvestrant | Group 2: Fulvestrant + Dasatinib | Group 3: Fulvestrant + MK-0646 | Group 4: Fulvestrant, MK-0646 + Dasatinib
Started | 2 | 3 | 1 | 0 (Zero participants started due to smaller sample size.)
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Fulvestrant | Group 2: Fulvestrant + Dasatinib | Group 3: Fulvestrant + MK-0646 | Group 4: Fulvestrant, MK-0646 + Dasatinib | Total
Number analyzed (Participants) | 2 | 3 | 1 | 0 | 6
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 2 | 2 | 1 |  | 5
  >=65 years | 0 | 1 | 0 |  | 1
Age, Continuous [Median (Full Range); unit: years] | 51 [40 to 62] | 63 [53 to 72] | 36 [36 to 36] |  | 57.5 [36 to 72]
Gender [Number; unit: participants]
  Female | 2 | 3 | 1 |  | 6
  Male | 0 | 0 | 0 |  | 0
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 1 |  | 2
  Not Hispanic or Latino | 2 | 2 | 0 |  | 4
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 1 | 0 | 0 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 |  | 0
  White | 1 | 3 | 1 |  | 5
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 1 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase I Maximum Tolerated Dose (MTD) for Dose Level 1
Description: Maximum Tolerated Dose (MTD) defined as the dose or dose-combination that has the mean posterior toxicity rate closest to the target toxicity rate of 0.33. Dose levels reviewed with each 28 day cycle. Treatment dose levels:
  Fulvestrant will be given using a loading dose of 500 mg intramuscularly (IM) on day 1 as two 250 mg/5 ml injections, followed by 500 mg IM on day 15 and on day 1 of each subsequent 28- day (+/- 2 days) cycle.
  MK-0646 will be given intravenously on days 1,8, 15, and 22 for each cycle at one of the two dose levels: 1) 5 mg/kg or 2) 10 mg/kg (Dose level 1)
  Dasatinib will be given orally (PO) continuously on days 1 -28 for each cycle at one of two dose levels: 1) 70 mg po daily or 2) 100 mg po daily
Time Frame: 28 day cycle
Population: Study terminated early; Analysis not available due to smaller sample size.
Arm/Group | Group 1: Fulvestrant | Group 2: Fulvestrant + Dasatinib | Group 3: Fulvestrant + MK-0646 | Group 4: Fulvestrant, MK-0646 + Dasatinib
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Patient Response (+ Time to Disease Progression)
Time Frame: Baseline, after two 28 day cycles, until disease progression.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event evaluation through each 28 day cycle and 3-4 weeks after the last cycle. Overall study collection period May 2010 to January 2012.
Arm/Group | Group 1: Fulvestrant | Group 2: Fulvestrant + Dasatinib | Group 3: Fulvestrant + MK-0646 | Group 4: Fulvestrant, MK-0646 + Dasatinib
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fulvestrant (N=2) | Group 2: Fulvestrant + Dasatinib (N=3) | Group 3: Fulvestrant + MK-0646 (N=1) | Group 4: Fulvestrant, MK-0646 + Dasatinib (N=0)
Gait abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fulvestrant (N=2) | Group 2: Fulvestrant + Dasatinib (N=3) | Group 3: Fulvestrant + MK-0646 (N=1) | Group 4: Fulvestrant, MK-0646 + Dasatinib (N=0)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (5) | 2 (8) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal Blood Tests (Blood and lymphatic system disorders) | 2 (4) | 3 (12) | 0 (0) | 0 (0) — Increase/Decreased White Blood Count (WBC), Absolute Neutrophil count (ANC), Hematocrit (HCT), Red Blood Cells (RBC)
Bone Pain, Generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte absolute count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Burning Sensation in throat (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash/Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Edema limbs (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 3 (4) | 1 (1) | 0 (0)
Fever (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Growth hormone abnormal (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Hot flashes (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic disorders (Metabolism and nutrition disorders) | 2 (12) | 3 (20) | 1 (9) | 0 (0) — Increased/Decreased Albumin, AST, BUN, Carbon Dioxide, Chloride Serum, HCT, RBC, WBC, Phosphorus Serum, Total Protein
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (3) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Paresthesia of the hand (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy, Leg (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Red irritated eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 2 (8) | 2 (6) | 1 (1) | 0 (0) — Body, Shoulder, Hip, Back, Arm, Leg, Heel.
Palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pressure Chest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum glucose decrease (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sweating (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No